CLINICAL TRIAL: NCT03365531
Title: A Randomized Controlled Trial of Caloric Restriction vs. Alternate-Day Fasting in Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: RCT of Caloric Restriction vs. Alternate-Day Fasting in Non-Alcoholic Fatty Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701956; OCR16250 (Other: University of Florida)
Record Dates: First submitted 2017-10-20; First posted 2017-12-07 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: NAFLD; Obesity; Diabetes Mellitus, Type 2
Keywords: fasting
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus, Type 2; Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial of Caloric Restriction vs. Alternate-Day Fasting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate Daily Fasting (ADF) (Experimental): Participants randomized to the ADF group will alternate between a day of ad lib feeding and a day of nearly no energy intake. Participants will be prescribed a core diet for feeding days that meets 110% of their estimated calorie needs within the fixed macronutrient distribution of 50% CHO, 20% PRO, and 30% FAT. In accordance with the ad lib feeding protocol, optional modules of similar macronutrient content will be prescribed, each providing an additional 200 kcals. Meal timing will not be restricted on these days. On fasting days, participants will be asked to consume 16 oz. of G2 Gatorade (40 kcal) in the morning and then only water or non-caloric beverages for the rest of the day.
  Interventions: Other: Alternate Daily Fasting (ADF)
- Caloric Restriction (Active Comparator): Participants randomized to the CR group will consume a diet of fixed energy designed to yield a 500 kcal/d deficit with a macronutrient distribution of 50% CHO, 20% PRO, and 30% FAT. Meal timing and caloric distribution will not be restricted.
  Interventions: Other: Caloric Restriction (CR)

INTERVENTIONS:
Other: Alternate Daily Fasting (ADF) — See ADF arm for details
  Arms: Alternate Daily Fasting (ADF)
Other: Caloric Restriction (CR) — See CR arm for details
  Arms: Caloric Restriction

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) in patients with diabetes (T2DM) is increasing in prevalence and can lead to cirrhosis. Lifestyle intervention with caloric restriction (CR) is the cornerstone of treatment but remission is variable. Alternatively, the PI has shown alternate day fasting (ADF) is safe and well tolerated in obese patients and there might be additional beneficial effects. The objective is to combine the expertise of the PI with this novel intervention and the expertise of Dr. Cusi in NAFLD to explore the effects of ADF vs CR in patients with NAFLD and T2DM to test the following hypotheses:

H1: In patients with NAFLD and T2DM, the ADF intervention will result in more favorable metabolic changes than CR:

H1a: Hepatic triglyceride by MRS will decrease more with ADF than CR (Primary Outcome) and remain lower following a period of free living H1b: There will be greater improvements in glucose homeostasis following ADF vs CR H1c: There will be greater improvement in lipid metabolism following ADF vs CR and changes in ketone metabolism will predict changes in hepatic triglyceride content H2: ADF will have similar safety and tolerability and result in a similar degree of weight loss in participants with NAFLD and DM compared to CR

DETAILED DESCRIPTION:
Rationale:

Non alcoholic fatty liver disease (NAFLD) has a prevalence of up to 80% in patients with T2DM and obesity and can lead to steatohepatitis (NASH) and fibrosis as well as cirrhosis and hepatocellular carcinoma. As NAFLD is associated with increased risk of cardiovascular disease and mortality and as NAFLD-induced liver disease is anticipated to be the most common indication for liver transplantation over the next decade, treatment options are desperately needed but very few are available.

Weight loss with caloric restriction (CR) is the preferred treatment of NAFLD, however successful maintenance of a significant weight loss is difficult to achieve. Additionally, despite significant association between degree of weight loss and improvements in NASH and NAFLD, there is extensive overlap in the response among populations. This suggests that it may not be weight loss in general, but rather the mechanistic underpinnings of the weight loss that potentiate the therapeutic effects. A study comparing dietary carbohydrate restriction vs CR in obese subjects with NAFLD found that, despite similar weight loss between groups, there was greater hepatic triglyceride reduction with carbohydrate restriction and this reduction was highly correlated with plasma ketone concentrations. Hence, although weight loss is ostensibly important, there might be additional factors beyond just weight loss per se causing the improvements in NASH. Therefore, rather than weight loss, reduction in intrahepatic triglyceride will be the primary endpoint of this proposal.

Progression to NASH and beyond is largely due to a spectrum of metabolic abnormalities including ectopic hepatic fat accumulation, insulin resistance, and abnormal lipid metabolism. A recent animal study showed blunted ketogenesis in NASH and suggested the overall etiology was due to inefficient oxidation and disposal of free fatty acids in the liver. A fasting paradigm, or facilitating times of ketosis that could then normalize lipid metabolism, might be one of the additional factors beyond weight loss that ensures improvements in NAFLD and NASH.

Intermittent fasting (IF) is a dietary intervention whereby food is restricted for varying timeframes, including alternate day fasting (ADF) where no or very few calories are given for a day or more with ad lib feeding in between. In animal models, IF has been shown to have numerous beneficial effects, many in excess of those seen with CR. In a mouse model of NAFLD, IF resulted in improvements in hepatic steatosis and inflammation along with gene expression changes showing enhanced activation of lipid oxidation and reduction of lipid synthesis. These benefits may be due to "flipping the metabolic switch" from glucose to ketone utilization for primary cellular energy needs. Data are only beginning to emerge on the effects of IF in humans, and very few studies have focused on ketone production as a mediator of positive outcomes. There are no data on the effect of ADF on NAFLD.

Specific Aims:

SA1: To compare the effect of ADF vs CR on metabolic changes including liver fat, glucose homeostasis, lipid metabolism, and inflammation in patients with NAFLD and T2DM SA1a: To determine changes in hepatic triglyceride by MRS after 4 weeks of ADF and after 4 weeks of ad lib diet SA1b: To determine changes in glucose homeostasis SA1c: To determine changes in whole body lipid metabolism and inflammation SA2: To determine the safety, tolerability, and effectiveness on weight loss of ADF vs CR SA2a: To determine safety of ADF SA2b: To compare changes in body weight, body composition, physical activity, physical functioning and physical fitness SA2c: To determine effect on eating behaviors, hunger/satiety, and body image SA2d: To determine effect on cognition and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patient must give study-specific informed consent on an IRB-approved consent prior to any research related procedures or study treatment.
* Patient must be at least 18 years at the time of consent Adenocarcinoma of the prostate with AJCC Clinical Stage T1to T3b disease with histological evaluation via biopsy or repeat biopsy within 12 months prior to registration. Refer to Appendix IV for clarification on study eligibility and AJCC stage group.
* Patients must undergo a pretreatment diagnostic MRI of the prostate on a 1.5T to 3T Tesla machine within 6 months prior to study registration.
* A focal IPT must be visible on MRI within the prostate and/or seminal vesicles and this MRI must be obtained within 6 months of planning CT scan.
* A biopsy of the dominant lesion is recommended but not required. If an ultrasound guided sextant biopsy was positive for prostatic adenocarcinoma in the area of the MRI identified intraprostatic lesion, this will be acceptable and another guided biopsy targeting the MRI identified disease will not be necessary.
* Patients with at least one of the following high-risk factors: cT3a-T3b OR Gleason 9-10 OR PSA > 30 OR more than 1 high-risk factors must be present: clinical stage of T3, Gleason score 8-10, or PSA 20 ng/ml or greater.
* Hemoglobin must be ≥ 10 g/ml within 4 months prior to registration.
* Zubrod performance status must be 0-1 within 4 months prior to registration.
* If patient has child-producing potential, they must be willing to use medically acceptable contraception during treatment and must be advised to use it for at least 1 year thereafter. This is not applicable if the patient is not sexually active or has had a vasectomy. Please document as such.
* Patients must be able to start treatment within 16 weeks of registration.

Exclusion Criteria:

* T4 prostate disease on CT, MRI, or physical exam.
* Patients unable to undergo MRI of the prostate.
* Patients with a greater than 25% change in prostate volume from the pretreatment MRI of the prostate demonstrating the IPT and the treatment planning MRI. Patients in this case must undergo a repeat diagnostic MRI on a 1.5T to 3.0T Tesla machine and an IPT must still be visible.
* IPT that is more than 75% of the prostate volume when measured on the CT simulation scan.
* Evidence of distant metastasis (M1).
* Patients with positive nodes on cross-sectional imaging.
* Previous prostate cancer local treatment including prostatectomy, hyperthermia, high intensity focused ultrasound, brachytherapy, external-beam radiation therapy, and/or cryotherapy.
* Prior pelvic radiation therapy.
* No prior myocardial infarction within the last 6 months, congestive heart failure, or end stage renal disease.
* Active inflammatory bowel disease (diverticulitis, Crohn's disease, ulcerative colitis) affecting the rectum.
* Bilateral hip replacement
* Prior intrapelvic surgery. This includes the following:Bladder surgery,Transrectal or rectal surgery other than prostate biopsy, Polypectomy or hemorrhoid removal or banding
* Prior transurethral resection of the prostate (TURP) or laser ablation for benign prostatic hyperplasia (BPH).
* Patients receiving continuous and current anticoagulation with warfarin sodium (Coumadin), heparin sodium, clopidogrel bisulfate (Plavix), dabigatran etexilate mesylate (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), edoxaban (Savaysa), enoxaparin sodium (Lovenox), prasugrel (Effient), ticagrelor (Brilinta), aspirin/er dipyridamole (Aggrenox), or fondaparinux sodium (Arixtra).
* Patients with posterior or posterolateral extracapsular extension of prostate cancer. If this is present, it must resolve on diagnostic MRI after 2 to 3 months of neoadjuvant androgen deprivation therapy prior to enrollment. Refer to Appendix V for definition of extracapsular extension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Hepatic Triglyceride by MRS | Baseline up to 8 weeks
  To determine changes in hepatic triglyceride by MRS after 4 weeks of ADF (Primary outcome) and after 4 weeks of ad lib diet

SECONDARY OUTCOMES:
Changes in Glucose Homeostasis | Baseline through 4 weeks
  To determine changes in glucose homeostasis as measured by: Overall and hepatic insulin sensitivity following OGTT using the Matusda index
Changes in whole body lipid metabolism - Adipose tissue insulin sensitivity by AdipoIR and fasting and postprandial free fatty acid excursion | Baseline through 4 weeks
  To determine changes in whole body lipid metabolism and inflammation as measured by: Adipose tissue insulin sensitivity by AdipoIR and fasting and postprandial free fatty acid excursion. Adipo-IR index (fasting, FFAs x insulin.
Safety of ADF -Liver Magnetic Resonance Spectroscopy (MRS) | Baseline through 4 weeks
  MRS to determine hepatic fat content and elasticity
Safety of ADF -Fibroscan. | Baseline through 4 weeks
  For liver steatosis (CAP) and fibrosis (VCTE) measurements
Safety of ADF - blood | Baseline through 4 weeks
  To determine safety of ADF measured by complete metabolic panel, glucose, ketones, and free fatty acids
To compare changes body composition measured | Baseline up to 8 weeks
  To compare changes in body weight, body composition measured by: Dual-energy x-ray absorptiometry (DEXA) to include weight
Effect on eating behaviors | Baseline up to 8 weeks
  Binge Eating Disorder Questionnaire: individuals can be categorized into three groups according to established cut-scores of binge eating severity. These groups are characterized by no binge eating (score ≤ 17), mild to moderate binge eating (score of 18 - 26) and severe binge eating (score ≥ 27)
Cognitive function | Baseline up to 8 weeks
  Effect on cognition and quality of life NIH Cognitive Toolbox
Diet Tolerability | Baseline up to 8 weeks
  ADF NAFLD Diet Tolerability a Likert scale design from 1-5, with 5 as strongly agree evaluating feasting days.

CONTACTS AND LOCATIONS:
Overall Officials: William T Donahoo, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Need to determine if able to de-identify enough relevant individual participant data to make sharing worthwhile and appropriate for this very small study.